CLINICAL TRIAL: NCT07058233
Title: Oral Nutritional Supplementation and Weight Changes During Therapy in Malnourished Patients With Resistant Tuberculosis: A Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSUP Persahabatan (Other)
Collaborators: Otsuka Holdings Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25/UN2.F1/ETIK/PPM.00.02/2022; Otsuka Holding (Other: Oral Nutritional Supplementation); Global Fund to Fight AIDS, TB (Other: Infection Disease)
Record Dates: First submitted 2025-06-19; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2022-12

CONDITIONS: Tuberculosis Multi Drug Resistant Active; Rifampin-Resistant Pulmonary Tuberculosis; Pre-xdr tb
Keywords: Drug-resistant tuberculosis; oral nutritional supplementation; malnutrition; total protein; globuline
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: one group intervention (standard treatment + Oral Nutritional Supplementation) and one group placebo (standard treatment only)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): standard Oral Nutritional Supplement (ONS) in the form of a soy-based drink (235 kcal/200mL: 10.34 g protein, 7.9 g fat, 30.61 g carbohydrate; Protein; Otsuka) with the instruction to consume three (3) sachets per day (total of 705 kcal and 31 grams of protein) plus standard treatment.
  Interventions: Dietary Supplement: Oral nutritional supplementation
- Control group (No Intervention): standard treatment only

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplementation — Oral Nutritional Supplement (ONS) in the form of a soy-based drink (235 kcal/200mL: 10.34 g protein, 7.9 g fat, 30.61 g carbohydrate; Protein)
  Arms: Intervention group

SUMMARY:
Tuberculosis increases energy demands and protein breakdown, leading to muscle wasting. Malnutrition and minimal weight gain less than 5% in first two months predict treatment failure. Malnutrition is defined as weight loss more than 5% in three months and Body Mass Index (BMI) ≤ 20 kg/m². This study assesses weight changes with high-energy, high-protein oral nutritional supplementation (ONS).

DETAILED DESCRIPTION:
Tuberculosis (TB) is linked to poverty, malnutrition, and reduced immunity, with malnutrition both contributing to and resulting from TB.1-3 Active TB increases energy needs, causes protein breakdown, and leads to muscle wasting. Malnutrition, which is common in TB patients, worsens clinical outcomes and increases the risk of death.1 TB treatments can also cause nausea and vomiting, further contributing to malnutrition.4 Thus integrated management is essential for successful treatment.

In India, 68.6% of MDR-TB patients without HIV infection are malnourished, a prevalence comparable to that observed among MDR-TB patients at Persahabatan General Hospital, Jakarta, Indonesia (51.8%).5,6 Malnourished MDR TB patients have worse clinical outcomes, more side effects, and a higher risk of death.7 A BMI under 18.5 kg/m2 and inadequate weight gain during treatment indicate a poor response and increased risk of recurrence.1 Failure to gain weight (≤ 5%) in the first two months of treatment has been demonstrated to be linked to TB recurrence.8 Oral nutritional supplements have demonstrated the potential to improve nutritional status, muscle strength, and immunity, thus potentially facilitating an accelerated treatment process. Studies have also shown that nutritional supplements can improve BMI and gamma interferon levels.9 However, some studies have indicated that despite increased macronutrient intake, MDR TB patients may still experience a decline in body weight.10 This study aims to evaluate whether oral nutritional supplements providing 705 kcal and 30.5 grams of protein daily during the first two months can increase body weight and improve other clinical outcomes of MDR TB patients, including the impact of supplementation on albumin, globulin, erythrocyte sedimentation rate (ESR), and C-reactive protein (CRP) levels.

ELIGIBILITY:
Inclusion Criteria:

* Who had access to electronic devices (e.g., mobile phones) for adherence monitoring
* individuals newly diagnosed with rifampicin-resistant pulmonary tuberculosis (RR-TB), multidrug-resistant tuberculosis (MDR-TB), or pre-extensively drug-resistant tuberculosis (Pre-XDR-TB) at the drug-resistant tuberculosis outpatient clinic of Persahabatan General Hospital, Jakarta, Indonesia.
* BMI of 13-20 kg/m²
* had received standardized or individualized treatment regimens for seven days
* had no severe drug-induced hepatitis indicated by elevated liver enzymes >5 times the normal upper limit

Exclusion Criteria:

* individuals with HIV infection,
* end-stage renal failure,
* severe anemia (hemoglobin <8 g/dL),
* severe hypoalbuminemia (albumin <2.5 g/dL),
* acute or chronic liver diseases (including hepatitis, cirrhosis, or jaundice),
* cancer,
* interstitial lung disease (ILD),
* anatomical gastrointestinal disorders (either congenital or post-surgical),
* diabetes mellitus,
* long-term corticosteroid or immunosuppressant therapy
* other acute pulmonary infections such as pneumonia,
* exacerbations of chronic obstructive pulmonary disease (COPD), or asthma

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Body weight | Pre intervention and post intervention (at 60 days)
  A change in body weight in kg

SECONDARY OUTCOMES:
Daily food intake | From enrollment to 60 days after enrollment
  Daily food intake of total energy, protein, fat, and carbohydrates. The subjects were given a form to record food intake 3 times a week (2 working days and 1 day off) for 8 weeks including the type and amount of food measured using standard units of spoons, glasses, etc. Furthermore, the intake data was converted into grams using a food ingredient analysis list and then analyzed using the 2007 nutrisurvey.
Albumin | Pre intervention and post intervention (at 60 days)
  Serum albumin is measured by taking peripheral venous blood samples with units of g/dL.
CRP | Pre intervention and post intervention (at 60 days)
  CRP is measured by taking peripheral venous blood samples in mg/dL units.
Total protein | Pre intervention and post intervention (at 60 days)
  Total protein is measured using a peripheral venous blood sample in g/dL units.
ESR | Pre intervention and post intervention (at 60 days)
  Erythrocyte sedimentation rate is measured using a peripheral venous blood sample in mm/hour units.

CONTACTS AND LOCATIONS:
Overall Officials: Fathiyah Isbaniah Sp.P(K), Dr., dr., Study Chair — Department of Pulmonology and Respiratory Medicine Faculty of Medicine, Universitas Indonesia, Persahabatan General Hospital, Jakarta
Locations (1):
- Rumah Sakit Umum Pusat Persahabatan, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No